CLINICAL TRIAL: NCT03917355
Title: Study of the Link Between Patient/Psychiatrist Motor Synchronization and Treatment Adhesion in Patients With First Psychotic Episode, ASMASS Project
Brief Title: Nonverbal Synchrony, Therapeutic Alliance and Treatment Engagement in First Episode Schizophrenia
Acronym: ASMASS
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0070
Record Dates: First submitted 2019-03-26; First posted 2019-04-17 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenics
MeSH Terms: interventions — Therapeutic Alliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Nonverbal synchrony, therapeutic alliance — Association between motor synchronisation in psychiatrist/patient dyad and patient therapeutic adherence in patients with a first psychotic episode will be measured, 6 months after the first post hospitalisation consultation, using video without sound. Nonverbal synchrony, therapeutic alliance and treatment will evaluated.In this purpose, videos of patients and psychiatrist will be made (for all patients included), and the images will be analyzed.

SUMMARY:
The quality of the therapeutic intervention in a first psychotic episode is a major challenge for quality and effectiveness of treatment. This project aims to better understand the mechanisms underlying the quality of communication between patient and psychiatrist, especially those related to non-verbal communication. Psychiatrist/patient interpersonal motor synchronization is a reliable index of therapeutic alliance and a predictor of psychotherapy effectiveness. This project aims to show a link between psychiatrist and patient motor synchrony and treatment adherence. This link could be explained by an association between therapeutic alliance and motor synchronization.

DETAILED DESCRIPTION:
Several studies have highlighted the utmost importance of initial medical and psychosocial support during a first psychotic episode. Recent research has shown that non-verbal communication and particularly interpersonal motor synchronization between the patient and his psychiatrist is a key factor in therapeutic alliance. However, such hypothesis have never been tested in terms of treatment adherence neither in a first psychotic episode, nor during a 6-month follow-up. By measuring the interpersonal motor synchronization between the patient and psychiatrist during a video recorded interview at inclusion, month-3 and month-6, the project aims to validate the hypothesis that a high level of interpersonal synchronization should be associated with a high level of therapeutic alliance. This therapeutic alliance being hypothesized as a mediator between synchronization and treatment adherence, the project should show for the first time in a first psychotic episode that the use of reliable and objective variables extracted from the analysis of the synchronization between psychiatrist and patient allows to predict the outcome of therapeutic and treatment alliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients after hospitalisation for a first psychotic episode (OMS criteria 1992)
* Patients fluent in French (spoken and written)
* Age ≥ 18 years and < 50 years
* signed informed consent
* participation noted in medical files.

Exclusion Criteria:

* Inpatients
* History of brain trauma
* History of neurological disease
* Current Electro-convulsive-treatment
* Drug abuse and dependence (except for tabacco and cannabis)
* Pregnant/breast feeding woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a first psychotic episode
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Scale of therapeutic compliance | Baseline
  This scale in French version (Fond et al. 2017), is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).
Scale of therapeutic compliance | 3 months
  This scale in French version (Fond et al. 2017), is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).
Scale of therapeutic compliance | 6 months
  This scale in French version (Fond et al. 2017), is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).

SECONDARY OUTCOMES:
Therapeutic alliance | Baseline
  It is a self-administered questionnaire with 11 items that measures the alliance perceived by a patient towards his or her doctor. The scale is a 4-point ordinal scale ("Yes, it is true" to "No, it is totally false"). It has been validated in French (Misdrahi et al., 2009) and is a valid tool for measuring therapeutic alliance in schizophrenia. It concerns the patient's feelings about the therapeutic alliance. The 4 Ordinal Point Alliance Scale consists of eleven clearly stated items and easy to understand.
Therapeutic alliance | 3 months
  It is a self-administered questionnaire with 11 items that measures the alliance perceived by a patient towards his or her doctor. The scale is a 4-point ordinal scale ("Yes, it is true" to "No, it is totally false"). It has been validated in French (Misdrahi et al., 2009) and is a valid tool for measuring therapeutic alliance in schizophrenia. It concerns the patient's feelings about the therapeutic alliance. The 4 Ordinal Point Alliance Scale consists of eleven clearly stated items and easy to understand.
Therapeutic alliance | 6 months
  It is a self-administered questionnaire with 11 items that measures the alliance perceived by a patient towards his or her doctor. The scale is a 4-point ordinal scale ("Yes, it is true" to "No, it is totally false"). It has been validated in French (Misdrahi et al., 2009) and is a valid tool for measuring therapeutic alliance in schizophrenia. It concerns the patient's feelings about the therapeutic alliance. The 4 Ordinal Point Alliance Scale consists of eleven clearly stated items and easy to understand.
Positive and Negative Symptom Scale | Baseline
  The PANSS (Kay et al., 1987) is a 30-item scale for measuring symptomatology specific to psychotic disorders, including schizophrenia. It has been validated in French (Lançon et al., 2000). It is a 7-point Likert scale that ranges from 1 (absent) to 7 (extremely present), giving a positive symptomatology score that ranges from 7 to 49, negative symptomatology (7 to 49), general psychopathology (16 to 112) and a total score (30 to 210).
Positive and Negative Symptom Scale | 3 months
  The PANSS (Kay et al., 1987) is a 30-item scale for measuring symptomatology specific to psychotic disorders, including schizophrenia. It has been validated in French (Lançon et al., 2000). It is a 7-point Likert scale that ranges from 1 (absent) to 7 (extremely present), giving a positive symptomatology score that ranges from 7 to 49, negative symptomatology (7 to 49), general psychopathology (16 to 112) and a total score (30 to 210).
Positive and Negative Symptom Scale | 6 months
  The PANSS (Kay et al., 1987) is a 30-item scale for measuring symptomatology specific to psychotic disorders, including schizophrenia. It has been validated in French (Lançon et al., 2000). It is a 7-point Likert scale that ranges from 1 (absent) to 7 (extremely present), giving a positive symptomatology score that ranges from 7 to 49, negative symptomatology (7 to 49), general psychopathology (16 to 112) and a total score (30 to 210).
Clinical Assessment Interview for Negative Symptoms | Baseline
  CAINS is a recently developed tool to evaluate the 2 dimensions of negative symptomatology highlighted in the literature, i.e. the motivation dimension and the decreased emotional expressivity dimension. It has been translated into French by our team (Raffard et al., currently under validation). It includes 13 items (9 for the motivation dimension and 4 for the expressivity dimension) evaluated during a semi-structured interview.
Clinical Assessment Interview for Negative Symptoms | 3 months
  CAINS is a recently developed tool to evaluate the 2 dimensions of negative symptomatology highlighted in the literature, i.e. the motivation dimension and the decreased emotional expressivity dimension. It has been translated into French by our team (Raffard et al., currently under validation). It includes 13 items (9 for the motivation dimension and 4 for the expressivity dimension) evaluated during a semi-structured interview.
Clinical Assessment Interview for Negative Symptoms | 6 months
  CAINS is a recently developed tool to evaluate the 2 dimensions of negative symptomatology highlighted in the literature, i.e. the motivation dimension and the decreased emotional expressivity dimension. It has been translated into French by our team (Raffard et al., currently under validation). It includes 13 items (9 for the motivation dimension and 4 for the expressivity dimension) evaluated during a semi-structured interview.
Functioning Remission of General Schizophrenia | Baseline
  The FROGS scale will be used to assess patient functioning. This questionnaire was developed, in French, according to the method of a consensus of experts, following a search in the main databases. This questionnaire has a good internal consistency (α=0.909) and good external validity (GFE score, r=0.56). The factor analysis identified 3 areas: "social functioning", "daily life", "treatment". The stability of the questionnaire was validated with a new evaluation at 1.5 years of patients and shows a good correlation of FROGS scores with other functioning evaluation scales. This questionnaire therefore has solid psychometric qualities. A total score is computed based on the sum of its 19 items ranging each from 1 (do not do) to 5 (do perfectly). The lower the score, the lower the functioning.
Functioning Remission of General Schizophrenia | 3 months
  The FROGS scale will be used to assess patient functioning. This questionnaire was developed, in French, according to the method of a consensus of experts, following a search in the main databases. This questionnaire has a good internal consistency (α=0.909) and good external validity (GFE score, r=0.56). The factor analysis identified 3 areas: "social functioning", "daily life", "treatment". The stability of the questionnaire was validated with a new evaluation at 1.5 years of patients and shows a good correlation of FROGS scores with other functioning evaluation scales. This questionnaire therefore has solid psychometric qualities. A total score is computed based on the sum of its 19 items ranging each from 1 (do not do) to 5 (do perfectly). The lower the score, the lower the functioning.
Functioning Remission of General Schizophrenia | 6 months
  The FROGS scale will be used to assess patient functioning. This questionnaire was developed, in French, according to the method of a consensus of experts, following a search in the main databases. This questionnaire has a good internal consistency (α=0.909) and good external validity (GFE score, r=0.56). The factor analysis identified 3 areas: "social functioning", "daily life", "treatment". The stability of the questionnaire was validated with a new evaluation at 1.5 years of patients and shows a good correlation of FROGS scores with other functioning evaluation scales. This questionnaire therefore has solid psychometric qualities. A total score is computed based on the sum of its 19 items ranging each from 1 (do not do) to 5 (do perfectly). The lower the score, the lower the functioning.
French National Adult Reading Test | Baseline
  The Premorbid IQ will be assessed by the French National Adult Reading Test (fNART) (McKinnon & Mulligan, 2005). Based on the ability to pronounce 40 words with irregular spelling (1 point per correct answer), this test provides an estimate of the subject's premorbid IQ.
French National Adult Reading Test | 3 months
  The Premorbid IQ will be assessed by the French National Adult Reading Test (fNART) (McKinnon & Mulligan, 2005). Based on the ability to pronounce 40 words with irregular spelling (1 point per correct answer), this test provides an estimate of the subject's premorbid IQ.
French National Adult Reading Test | 6 months
  The Premorbid IQ will be assessed by the French National Adult Reading Test (fNART) (McKinnon & Mulligan, 2005). Based on the ability to pronounce 40 words with irregular spelling (1 point per correct answer), this test provides an estimate of the subject's premorbid IQ.
California Verbal Learning Test | Baseline
  The experimenter reads a list of 16 words. The patient must then return as many words as possible (immediate free recall), repeated 5 times. The experimenter reads a new list of 16 words, this new list serves as an interference. The patient is asked to return as many words as possible from the second list (immediate free recall). Then the patient is instructed to try to return as many words as possible from first list (free short term recall), then comes an indication phase. 20 minutes break without verbal tests. The patient is instructed again to return as many words as possible from first list (free long-term recall) and arrives to complete a new phase of indication (long-term indexed recall). This test highlights long-term memory recovery processes as well as long-term memory consolidation processes. The standard score is the Total Recall Responses (160).
California Verbal Learning Test | 3 months
  The experimenter reads a list of 16 words. The patient must then return as many words as possible (immediate free recall), repeated 5 times. The experimenter reads a new list of 16 words, this new list serves as an interference. The patient is asked to return as many words as possible from the second list (immediate free recall). Then the patient is instructed to try to return as many words as possible from first list (free short term recall), then comes an indication phase. 20 minutes break without verbal tests. The patient is instructed again to return as many words as possible from first list (free long-term recall) and arrives to complete a new phase of indication (long-term indexed recall). This test highlights long-term memory recovery processes as well as long-term memory consolidation processes. The standard score is the Total Recall Responses (160).
California Verbal Learning Test | 6 months
  The experimenter reads a list of 16 words. The patient must then return as many words as possible (immediate free recall), repeated 5 times. The experimenter reads a new list of 16 words, this new list serves as an interference. The patient is asked to return as many words as possible from the second list (immediate free recall). Then the patient is instructed to try to return as many words as possible from first list (free short term recall), then comes an indication phase. 20 minutes break without verbal tests. The patient is instructed again to return as many words as possible from first list (free long-term recall) and arrives to complete a new phase of indication (long-term indexed recall). This test highlights long-term memory recovery processes as well as long-term memory consolidation processes. The standard score is the Total Recall Responses (160).
Trail Making Test | Baseline
  This test is used to evaluate executive functions and more particularly mental flexibility. It is a timed test, with five conditions: visual exploration (condition 1), number order (condition 2), letter order (condition 3), number-letter flexibility (condition 4) and motor speed (condition 5). The main dependent variable to note is the difference in time between condition 4 - condition 1.
Trail Making Test | 3 months
  This test is used to evaluate executive functions and more particularly mental flexibility. It is a timed test, with five conditions: visual exploration (condition 1), number order (condition 2), letter order (condition 3), number-letter flexibility (condition 4) and motor speed (condition 5). The main dependent variable to note is the difference in time between condition 4 - condition 1.
Trail Making Test | 6 months
  This test is used to evaluate executive functions and more particularly mental flexibility. It is a timed test, with five conditions: visual exploration (condition 1), number order (condition 2), letter order (condition 3), number-letter flexibility (condition 4) and motor speed (condition 5). The main dependent variable to note is the difference in time between condition 4 - condition 1.
Energy Motion Analysis | Baseline
  Motion Energy Analysis is a valid, robust and objective measure of the degree of Motor Synchrony between two people.It is captured using two cameras oriented respectively towards the patient and the clinician. This video analysis consists in extracting the amount of movement present between two successive images (Number of pixels that differs between two successive video frames) and thus automatically extracting the activity of the patient and that of the clinician during an interview. The comparison between these two time series by cross-correlation gives a single measure r representing the quantity of Motor Synchrony present in the exchange between the patient and the clinician. Therefore MS ranges from 0 (no synchrony) to 1 (perfect synchrony).The higher the value, the higher the synchronisation.
Energy Motion Analysis | 3 months
  Motion Energy Analysis is a valid, robust and objective measure of the degree of Motor Synchrony between two people.It is captured using two cameras oriented respectively towards the patient and the clinician. This video analysis consists in extracting the amount of movement present between two successive images (Number of pixels that differs between two successive video frames) and thus automatically extracting the activity of the patient and that of the clinician during an interview. The comparison between these two time series by cross-correlation gives a single measure r representing the quantity of Motor Synchrony present in the exchange between the patient and the clinician. Therefore MS ranges from 0 (no synchrony) to 1 (perfect synchrony).The higher the value, the higher the synchronisation.
Energy Motion Analysis | 6 months
  Motion Energy Analysis is a valid, robust and objective measure of the degree of Motor Synchrony between two people.It is captured using two cameras oriented respectively towards the patient and the clinician. This video analysis consists in extracting the amount of movement present between two successive images (Number of pixels that differs between two successive video frames) and thus automatically extracting the activity of the patient and that of the clinician during an interview. The comparison between these two time series by cross-correlation gives a single measure r representing the quantity of Motor Synchrony present in the exchange between the patient and the clinician. Therefore MS ranges from 0 (no synchrony) to 1 (perfect synchrony).The higher the value, the higher the synchronisation.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No